CLINICAL TRIAL: NCT03601000
Title: Efficacy Study of Yi-Zhi-An-Shen Granules For Older Adults With Amnestic Mild Cognitive Impairment: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy Study of Yi-Zhi-An-Shen Granules For Older Adults With Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChengduUTCM-WWB-201801
Record Dates: First submitted 2018-04-05; First posted 2018-07-26 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Dysfunction
Keywords: amnestic
MeSH Terms: conditions — Cognitive Dysfunction | interventions — yi-zhi-an-shen

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yi-Zhi-An-Shen (Experimental): Yi-Zhi-An-Shen Granules given three times every day for 16 weeks.
  Interventions: Drug: Yi-Zhi-An-Shen
- Placebo (Placebo Comparator): Placebo given three times every day for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yi-Zhi-An-Shen — Yi-Zhi-An-Shen Granules 5g given three times a day for up to 16 weeks.
  Arms: Yi-Zhi-An-Shen
Drug: Placebo — Placebo granules 5g given three times a day for up to 16 weeks.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the safety and efficacy of Yi-Zhi-An-Shen Granules in participants with amnestic mild cognitive impairment (aMCI).

DETAILED DESCRIPTION:
The investigators performed a randomized, placebo-controlled, double-blind study on evaluating effect of Yi-Zhi-An-Shen Granules on cognition, sleep quality, and gut microbiome of older adults with amnestic mild cognitive impairment (aMCI). The investigators plan to involve 80 cases for observation in 2 years (40 cases for each group), expecting that cognition and sleep quality of aMCI patients can be improved by Yi-Zhi-An-Shen Granules versus placebo, and discussing the differences between individuals with aMCI and ones with normal cognition, also investigating whether this Chinese medicine compound can regulate gut microbiome of older individuals with aMCI.

ELIGIBILITY:
Inclusion Criteria:

* Subject has assigned informed consent to participate in the study and continues to give willing consent for participation
* Age from 60 to 85 years with a diagnosis of aMCI
* Educational level of at least 6 years
* Availability of a "study partner" who can assist in completing rating scales for the duration of the study
* Cognitive complaints reported by the subject and confirmed by the "study partner"
* Clinical Dementia Rating (CDR) global score of 0.5, and memory item score of 0.5
* Mini-mental state examination (MMSE) score of 24-30
* Diagnostic and Statistical Manual of Mental Disorders, Version 5 (DSM-V) criteria of dementia not fulfilled

Exclusion Criteria:

* Has been previously enrolled in this study and received the investigational product
* Has received an investigational product within 30 days prior to screening
* Has received disease-modifying therapy
* Has a known allergy to the study drug or any of its constituents
* Has a history of alcohol abuse or alcohol dependency in the 3 years prior to study entry, or is an alcoholic or drug addict, as determined by the investigator
* Has ongoing clinically significant (as judged by the investigator), metabolic or any other disease that could currently cause impaired memory (e.g., untreated thyroid disease, vitamin or other nutritional deficiencies, chronic kidney, or liver disease)
* Memory impairment that can be attributed to a disease or condition other than an early phase neurodegenerative syndrome
* Has a parkinsonian movement disorder
* Use of psychoactive medications that would affect the subject's ability to reliably perform neurocognitive testing or create uncertainty in distinguishing between the effects of the psychoactive medication and the subject's underlying cognitive impairment (e.g., benzodiazepines, sedatives, antipsychotics)
* History of major recurrent depressive disorder (DSM-V) within the last 5 years prior to screening
* Has a brain tumor or other intracranial lesion, a disturbance of cerebral spinal fluid circulation (e.g., normal pressure hydrocephalus), and/or a significant history of head trauma or brain surgery
* Has signs of major cerebrovascular disease, with score of modified Hachinski Ischemia Score (mHIS) at more than 4, or as verified by medical history and/or brain MRI or CT
* Has severe visual or hearing impairments that cannot cooperate with examinations
* Has severe digestive system diseases
* Has received antibiotics within 60 days prior to screening

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Alzheimer´s Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Score | Baseline, 16 weeks, 22 months
  The ADAS-Cog was developed as an outcome measure for global cognition in clinical trials. The ADAS-Cog assesses multiple cognitive domains including memory, language, praxis, and orientation, for a total of 70 points (0: no cognitive impairment; 70: severe impairment). An improvement of 4 points is used as a criterion of clinically effective anti-dementia drugs.

SECONDARY OUTCOMES:
Change from Baseline in the Mini Mental Status Examination (MMSE) | Baseline, 8 weeks, 16 weeks, 10 months, 16 months, 22 months
  Changes in the global cognitive function will be accessed by MMSE to evaluate the severity of subjects' cognitive impairment. The MMSE includes orientation, registration, attention and calculation, recalling and language tests, for a total of 30 points. A score below 24 is considered abnormal for dementia screening.
Change from Baseline in the Montreal Cognitive Assessment (MoCA) | Baseline, 8 weeks, 16 weeks, 10 months, 16 months, 22 months
  MoCA (Changsha Version), as a assessment tool for rapid MCI screening, will be used to assess changes in the global cognitive function. With a total of 30 points, a score below 25 is considered abnormal, and the lower score indicates the worse cognition.
Change from Baseline in the Clinical Dementia Rating Scale (CDR) | Baseline, 16 weeks, 22 months
  The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to AD and related dementias: Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care. Scores on the CDR range from 0 (no impairment) to 3 (severe impairment). The total CDR ratings for each of the six cognitive/functional domains can be added to create a CDR sum of boxes (CDR-SB).
Change from Baseline in the Activity of Daily Living (ADL) | Baseline, 8 weeks, 16 weeks, 10 months, 16 months, 22 months
  ADLs will be assessed including basic activities of daily living (BADL) and instrumental activities of daily living (IADL). An individual's BADL will be evaluated mainly by the subjects' performance from the perspectives of bathing, dressing, grooming, initiation, toileting and feeding, with six items and a sum of scores ranging from 0 (normal) to 24 (complete dependence on others). And modified Lawton Instrumental Activities of Daily Living Scale will be used to measure the IADL of a subject, with eight items and a sum of scores ranging from 0 (normal) to 32 (complete dependence on others).
Change from Baseline in the Pittsburgh sleep quality index (PSQI) | Baseline, 8 weeks, 16 weeks, 10 months, 16 months, 22 months
  The PSQI will be used to assess participants' comprehensive sleep quality, including sleep quality, sleep duration, sleep efficiency, sleep disorders, daytime dysfunction, sleeping aids, etc. The total score is 21, with a higher score indicating a worse sleep quality.
Differences between patients with aMCI and individuals with normal cognition in gut microbiome. | Baseline, 16 Weeks
  The investigators will collect some fecal samples from participants. Then, differences in gut microbiome between patients with aMCI and individuals with normal cognition will be analyzed using 16SrDNA and Metagenomics analyses. When it is available, the investigators will also assess the change in gut microbiome between the treatment group and the placebo group after the intervention of YZASG.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wu, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Teaching Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Welfare Institution of Emei Civil Administration, Leshan, Sichuan

REFERENCES:
- [Background] Miao YC, Tian JZ, Shi J, Mao M. Effects of Chinese medicine for tonifying the kidney and resolving phlegm and blood stasis in treating patients with amnestic mild cognitive impairment: a randomized, double-blind and parallel-controlled trial. Zhong Xi Yi Jie He Xue Bao. 2012 Apr;10(4):390-7. doi: 10.3736/jcim20120407. PMID 22500712
- [Derived] Yue S, He T, Li B, Qu Y, Peng H, Chen J, Lei M, Chen C, Wu W. Effectiveness of Yi-Zhi-An-Shen granules on cognition and sleep quality in older adults with amnestic mild cognitive impairment: protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2019 Aug 20;20(1):518. doi: 10.1186/s13063-019-3607-x. PMID 31429790

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT03601000/Prot_SAP_000.pdf